CLINICAL TRIAL: NCT06336980
Title: Creating Welcoming Faith Communities for Believers With Serious Mental Illnesses: Testing an Environmental, Behavior-Oriented Intervention
Brief Title: Creating Welcoming Faith Communities for People With Serious Mental Illnesses
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Temple University (Other)
Collaborators: National Institute on Disability, Independent Living, and Rehabilitation Research (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 31021
Record Dates: First submitted 2024-02-27; First posted 2024-03-29 (Actual); Last update posted 2024-05-06 (Actual); Status verified 2024-05

CONDITIONS: Other
Keywords: inclusion; stigma reduction; faith communities

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Behavior intervention to increase inclusionary practices (Experimental): Each congregation will participate in the intervention for 11-12 months
  Interventions: Behavioral: Increasing Inclusionary Practices in Faith Communities

INTERVENTIONS:
Behavioral: Increasing Inclusionary Practices in Faith Communities — Congregational inclusion committees will participate in monthly training meetings for approximately 1 year. Each month a new inclusion practice will be introduced and then the committee will be asked to implement it in their congregation. The 11 practice areas are:1) assessing inclusion needs of members, 2) providing opportunities for members with serious mental illness (SMI) to take on roles and responsibilities, 3) creating an inclusion committee, 4) ensuring that members with SMI are welcomed to all events, 5) creating sensory friendly spaces, 6) offer participation opportunities in multiple formats, 7) adopt policies and practices to support inclusion, 8) using inclusive language, 9) ensure that external communications indicate the congregation is welcoming to all, 10) providing support to family members of individuals with SMI, and 11) conducing outreach to mental health support systems. Goals may vary per congregation based on their current practices, needs, and preferences.

SUMMARY:
The goal of this intervention study is to test a behavioral intervention to increase inclusionary practices toward individuals with serious mental illness in faith communities. The main questions it aims to answer are:

1. To determine if the behavior-based intervention leads to an increase in inclusionary practices (e.g., conducting outreach with mental health agencies).
2. To determine if the behavior-based intervention is effective in increasing inclusive practices by members and leaders of faith communities.
3. To determine if the intervention leads to a greater understand of mental illness and a decrease in stigmatizing beliefs by congregation members.
4. To determine if the intervention results in individuals with serious mental illness and their family members reporting less discrimination and increased inclusion.

Congregations will be asked to create an inclusion committee that will then work on developing systems and changing congregational practices to become more inclusive. All congregation members will be invited to a half-day training that will provide information on mental illness and inclusion, and will provide tips and strategies when they encounter situations or behaviors that are less familiar to them. All congregation members will be given the opportunity to participate in a survey about congregational practices.

ELIGIBILITY:
Inclusion Criteria:

* member or attendee of the faith community participating in the training

Exclusion Criteria:

* under the age of 18

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 700 (Estimated)
Dates: Start 2024-01-22 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Inclusionary practices | Will be measured once per month for the duration of the study up to one year.
  Researchers will evaluate inclusionary practices done in the congregation (e.g. create an intake form for new members). There might be up to 50 different practices. The number of practices will vary by congregation. Each practice will measured as being done or not (yes or no). A greater number of "yes" responses will indicate greater inclusionary practices.
Indicators of Welcome | Survey will be administered 2 times at the baseline and 11-12 months later at the end of the study
  These questions are only being given to everyone who took the survey including those who report they do not have a mental illness, those that report that they do, and those that report that they have a family member with a mental illness. There are 32 statements related to organizational processes and respondent experiences with inclusion in their congregation. There are an additional three statements specifically for those with family members with mental illness. The response options are yes, no, and I don't know. A greater number of "yes" responses would indicate a greater number of inclusionary practices and greater inclusive experiences and "no" or "I don't know" would indicate the opposite.
Mental Health Knowledge Questionnaire | Survey will be administered 2 times at the baseline and 11-12 months later at the end of the study
  These questions are only being given to participants who report that they do not mental illness. It consists of 6 statements related to knowledge about treatments and outcomes for individuals with mental illness. Response options range from strongly agree (6) to strongly disagree (1) on a 6-point scale. Stronger agreement or higher scores across statements indicates a higher level of knowledge about mental illness and a stronger disagreement or lower scores indicates less knowledge about mental illness.
Social Distance Scale | Survey will be administered 2 times at the baseline and 11-12 months later at the end of the study
  These questions are only being given to participants who report that they do not mental illness. This measure assesses participants's comfort level in being around people with mental illness. It was modified to include measures directly related to faith communities (e.g., would you feel comfortable having someone with a serious mental illness as a member of your congregation). There are 7 questions with response options that vary from strongly disagree (1) to strongly agree (6) on a 6-point scale. Stronger agreement or higher scores indicate a higher level of comfort with people with mental illness and stronger disagreement or lower scores indicate a lower level of comfort with people with mental illness.
Community Attitudes Toward the Mentally Ill | Survey will be administered 2 times at the baseline and 11-12 months later at the end of the study
  These questions are only being given to participants who report that they do not mental illness. There are 4 statements related to attitudes toward people with mental illness from this measure. The response options for each statement range from strongly disagree (1) to strongly agree (6) on a 6-point scale. Stronger agreement or higher scores across all questions indicate more negative attitudes toward those with mentally illness and stronger disagreement or lower scores (1) across all questions indicates more positive attitudes toward those with mental illness.
Reported and Intended Behavior Scale | Survey will be administered 2 times at the baseline and 11-12 months later at the end of the study
  These questions are only being given to participants who report that they do not mental illness. The measure is divided into two parts. The first 4 questions ask about the participants current experiences with people with mental illness. Response options include "yes" or "no, or not that I know of". A greater number of yes responses indicates more experience with individuals with mental illness. The second part includes 4 questions asking about a person's willingness to include people with mental illnesses in their life. The response options are from strongly disagree (1) to strongly agree (6) on a 6-point scale with stronger agreement or higher scores on each question indicating a greater willingness to associate with or include or have people with mental illnesses in their life in the future. Stronger disagreement or lower scores across questions indicates less willingness to associate with or include people with mental illnesses in their lives.
Sense of Belonging Scale | Survey will be administered 2 times at the baseline and 11-12 months later at the end of the study
  These 10 questions are only being given to participants who report having a mental illness or a family member with a mental illness. The questions ask participants the degree to which they feel welcomed and that they belong in a given environment. For this study that environment was their congregation. Response options range from strongly agree to strongly disagree on a 6-point scale. Stronger agreement or higher scores (6) on questions 2, 3, 4, 7, 8, 9 , and 10 and stronger disagreement (1) or lower scores on questions 1, 5, and 6 indicate a greater sense of belonging. Stronger disagreement (1) or lower scores to questions 2, 3, 4, 7, 8, 9, and 10 and stronger agreement (6) or higher scores to questions 1, 5, and 6 indicate less of a sense of belonging.

SECONDARY OUTCOMES:
University of California Los Angeles Loneliness Scale | Survey will be administered 2 times at the baseline and 11-12 months later at the end of the study
  These 3 questions are only being given to participants who report having a mental illness. The questions related to how often participants feel socially isolated or lonely. Response options range from 1) hardly ever, 2) some of the time, and 3) often. Responses (3) indicate increased loneliness and more "hardly ever" responses indicate less loneliness.
Lerman Quality of Life Interview | Survey will be administered 2 times at the baseline and 11-12 months later at the end of the study
  This measure is only presented to people who report having a mental illness. Only the first question from this scale is being asked as it correlates well to other items on the interview related to overall quality of life. The one question asks participants "how do you feel about your life in general?" Response options vary from terrible to delighted on a 7-point scale. Responses closer to 7 (delighted) indicate greater perceived quality of life and responses closer to 1 (terrible) indicate lower perceived quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- Temple Univeristy, Philadelphia, Pennsylvania, United States